CLINICAL TRIAL: NCT06999655
Title: Radicle EnergyTM 24_VKG: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Fatigue and Related Health Outcomes
Brief Title: Radicle Energy: A Study Assessing the Impact of Health and Wellness Products on Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2404_VKG
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-07

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their assigned sex at birth and health outcome score during enrollment, then randomized to one of the study arms. Each participant will have an equal chance of being assigned to any study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Control (Placebo Comparator): Energy Product Control
  Interventions: Dietary Supplement: Energy Placebo Control
- Active Product 1 (Experimental): Energy Active Product 1
  Interventions: Dietary Supplement: Energy Active Product 1
- Active Product 2 (Experimental): Energy Active Product 2
  Interventions: Dietary Supplement: Energy Active Product 2

INTERVENTIONS:
Dietary Supplement: Energy Placebo Control — Participants will use their Energy Placebo Control as directed for a period of 6 weeks.
  Arms: Placebo Control
Dietary Supplement: Energy Active Product 1 — Participants will use their Energy Active Product 1 as directed for a period of 6 weeks.
  Arms: Active Product 1
Dietary Supplement: Energy Active Product 2 — Participants will use their Energy Active Product 2 as directed for a period of 6 weeks.
  Arms: Active Product 2

SUMMARY:
A randomized, double-blind, placebo-controlled study assessing the impact of health and wellness products on fatigue and related health outcomes

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (2) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities

o Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed

* Resides in the United States
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

Report being pregnant, trying to become pregnant, or breastfeeding

* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  o NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

  o Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products and/or pose a safety risk
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue | 7 weeks
  Difference between rates of change over time in fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 8A (scale 8-40; where the higher scores correspond to more fatigue)

SECONDARY OUTCOMES:
Change in Cognitive Function | 7 weeks
  Difference between rates of change over time in cognitive function score as assessed by Patient Reported Outcome Measurement System (PROMIS) Cognitive Function 4A (scale 4-20; where the higher scores correspond to greater cognitive function)
Change in Sleep Disturbance | 7 weeks
  Difference between rates of change over time in sleep disturbance score as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance 4A (scale 4-20; where the higher scores correspond to more sleep disturbance)
Change in mood | 7 weeks
  Difference between rates of change over time in mood score as assessed by Patient Reported Outcome Measurement System (PROMIS) Depression 4A (scale 4-20; where the higher scores correspond to more feelings of depression)

OTHER OUTCOMES:
Minimal clinical importance difference (MCID) in fatigue | 7 weeks
  Likelihood of achieving a MCID in fatigue, as measured by PROMIS Fatigue 8A (scale 8-40; where the higher scores correspond to greater fatigue)
Minimal clinical importance difference (MCID) in cognitive function | 7 weeks
  Likelihood of achieving a MCID in cognitive function, as measured by PROMIS Cognitive Function Short Form 4A (scale 4-20; where the higher scores correspond to greater cognitive function)
Minimal clinical importance difference (MCID) in sleep disturbance | 7 weeks
  Likelihood of achieving a MCID in sleep disturbance, as measured by PROMIS Sleep Disturbance 4A (scale 4-20; where the higher scores correspond to greater sleep disturbance)
Minimal clinical importance difference (MCID) in mood | 7 weeks
  Likelihood of achieving a MCID in mood, as measured by PROMIS Depression 4A (scale 4-20; where the higher scores correspond to greater feelings of depression)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com